CLINICAL TRIAL: NCT02271295
Title: Impact on Morbidity and Mortality of Prophylactic Dosing of Low Molecular Weight Heparin in Child-Pugh B Cirrhotic Patients: a Randomized Controlled Study
Brief Title: Impact on Morbidity and Mortality of Prophylactic Dosing of Low Molecular Heparin in Child-Pugh B Cirrhotic Patients
Acronym: Childbenox
Status: Suspended | Phase: Phase 3 | Type: Interventional
Why Stopped: Premature discontinuation of inclusions by the sponsor for low inclusion
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P130926; AOM 13606 (Other Grant/Funding Number: Ministry of Health)
Record Dates: First submitted 2014-10-20; First posted 2014-10-22 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Cirrhosis
Keywords: Cirrhosis; Child B; decompensation; mortality; portal thrombosis; anticoagulation
MeSH Terms: conditions — Fibrosis | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enoxaparine (Experimental): 69 Child Pugh B7-C10, cirrhotic patients receiving anticoagulation treatment (daily subcutaneous injection of enoxaparin 4000UI/day) during 24 months
  Interventions: Drug: Enoxaparine
- Control (No Intervention): 69 Child Pugh B7-C10, cirrhotic patients not receiving anticoagulation treatment

INTERVENTIONS:
Drug: Enoxaparine — Enoxaparine 4000UI/day during 24 months
  Other Names: LOVENOX® 4000UI/day
  Arms: Enoxaparine

SUMMARY:
Thrombosis occurring in the small intrahepatic, as well as in the large vessels is involved in the progression of cirrhosis. Anticoagulation could reduce morbidity and mortality in cirrhotic patients

DETAILED DESCRIPTION:
Cirrhosis is the end-stage of all chronic liver diseases. Cirrhosis is a critical step in the natural history of liver disease, as it is associated with the occurrence of complications (so-called decompensation) and death. Life expectancy varies from 12-14 years in patients with compensated cirrhosis, to 2-4 years after decompensation.

Cirrhosis is associated with thrombosis of the intrahepatic portal and hepatic venous systems leading to parenchymal extinction (atrophy), liver dysfunction and portal hypertension. Regeneration in the areas without microthrombosis, and inflammation are powerful factors inducing liver cancer. Portal and hepatic venous thrombosis have been shown to participate in remodeling the liver architecture and are associated with a worsening outcome. Thrombosis in cirrhosis is thought to result from a procoagulant state due to an imbalance between pro and anticoagulant factor plasma levels, inflammation in and around blood vessels, and a marked slowing down of venous blood flow. Heparin administration, in animal models of liver fibrosis, decreases extra cellular matrix protein synthesis and fibrous tissue deposition. Recently, a reduction in liver decompensation and mortality has been shown in Child-Pugh B7-C10 cirrhotic patients assigned to receive a low dose of enoxaparin (4000IU/d), a low molecular weight heparin, for 48 weeks, compared to patients receiving no anticoagulation therapy.

These results are in line with the hypothesis of a protective role of anticoagulation in liver disease progression and a strong association between thrombosis and liver fibrosis.

So the main objective of the study is to compare the effect of a 2-year low dosing of Enoxaparin (4000 IU/day) versus no treatment on morbidity and mortality in patients with Child B7-C10 cirrhosis.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤75 years old
* A diagnosis of cirrhosis based on liver biopsy or on the combination of clinical, laboratory and imaging criteria
* Compensated Child-Pugh B7-C10
* Any of the following causal factors : past but controlled excessive alcohol intake (<30g/d for men and <20g/d for women), HCV infection without viral replication, HBV infection without viral replication on therapy, metabolic syndrome, biliary cirrhosis, auto-immune cirrhosis, hemochromatosis, cryptogenetic cirrhosis

Exclusion Criteria:

* Ascites, portal hypertensive bleeding or encephalopathy within the last 3 months prior to enrolment
* Hepatocellular carcinoma non considered in remission
* Budd Chiari syndrome non considered in remission
* Liver transplantation
* F2 or F3 varices without treatment in accordance with recommended guidelines (B-blockers, ligation or both)
* Portal vein thrombosis
* Transjugular intrahepatic portosystemic shunt
* Known extra-hepatic malignancies
* PT<35%
* Platelet count<50,000/mm3
* Haemoglobin level < 9g/dl
* Serum Albumin < 20g/L
* A bone mineral density T score of less than -4.0 at the lumbar spine or total hip
* Known HIV infection
* Ongoing anticoagulation or antiaggregation
* Renal insufficiency defined by creatinine clearance<60ml/mn
* Conditions at risk for spontaneous bleeding (except for portal hypertension) or hemostatic abnormalities not related to cirrhosis
* Pregnancy or breast-feeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-07-27 (Actual); Primary Completion 2019-07-02 (Estimated); Study Completion 2019-07-02 (Estimated)

PRIMARY OUTCOMES:
Morbidity and mortality at 24 months | 24 months
  To compare the effect of a 2-year low dosing of Enoxaparin (4000 IU/day) versus no treatment on morbidity and mortality in patients with Child B7-C10 cirrhosis.

SECONDARY OUTCOMES:
Mortality liver-related or not at 24 months | 24 months
  Two year overall survival and two year liver related survival considering non-liver death as a competive event.
Adverse events at 24 months | 24 months
  percentage of bleeding episodes not reported to portal hypertension, percentage of heparin induced thrombocytopenia, variation of bone mineral density (M24-M0/M0) and percentage of occurrence of osteoporosis at dual energy X-ray absorptiometry
Liver function and fibrosis at 24 months | 24 months
  * Variation of liver function tests (M24-M0/M0): PT, albumin and T bilirubin levels, Child-Pugh and MELD score
  * Variation of non-invasive tests of liver fibrosis (M24-M0/M0): fibrometer and cirrhometer scores, liver stiffness measurement using transient elastography.
Thrombosis at 24 months | 24 months
  Occurrence of portal vein (PV) thrombosis at Doppler ultrasound evaluation performed every 3 months or CT scan performed at M-1 and M24 (appendix 2) or hepatocellular carcinoma at Doppler ultrasound evaluation performed every 3 months or CT scan performed at M-1 and M24 and confirmed according to EASL recommendations
Compliance | 24 months
  record of unused packaging and information about compliance in a patient diary
Survival rate without completion | 30 months
  Survival rate without complication 6 months after completion of treatment as well as variation of liver function and portal hypertension parameters, occurrence of PV thrombosis, occurrence of bacterial infections
Portal hypertension parameters | 24 months
  Variation of portal hypertension parameters (M24-M0/M0): platelets count, esophageal varices size at endoscopic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Armelle Poujol-Robert, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hôpital Saint Antoine, Paris, France